CLINICAL TRIAL: NCT06715774
Title: Impact of Twin Block and Motion Class II Appliances on Hyoid Bone Position - A Retrospective Clinical Study
Acronym: Hyoid bone
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Romane Gilbert, University of Salamanca
Other Study IDs: RG-2024-ortho
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Hyoid Bone
Keywords: Hyoid bone, twin block, motion,

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Impact of Twin Block and Motion above Hyoid bone — All patients were submitted to preoperative and postoperative lateral teleradiography (Vatech D052SB, Puteaux, France), with the following exposure parameters: 75KV, Intensity10mA, exposition times 11s28, 112,8 mAs, using the Frankfort plane as reference parallel to the floor; moreover, patients were required to avoid moving and swallowing. Afterwards, digital datasets were uploaded and aligned into a digital therapeutic planning software (Orthalis®, Orqualceph®,group orqual) to accurately record the position changes of the hyoid bone at horizontal, vertical, and angular level, according the gender, facial biotype and airway complex, by measuring the following anatomical references:

SUMMARY:
Analyse the impact Twin block appliance and Motion on Hyoid Bone

DETAILED DESCRIPTION:
Patients were selected, divided en two homogenous groups and underwent preoperative and postoperative lateral teleradiograph scans. The datasets were subsequently uploaded into a digital treatment planning software to record the position changes of the hyoid bone at horizontal, vertical, angular, and airway complex level; additionally, the effect of gender, age at onset, treatment time, biotype, and their interactions with the group, have been also statistically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 10 and 16 years old, with sketelal class II, a ANB angle ≥4° according to the Steiner cephalometric analysis, with Twin block or Motion appliance

Exclusion Criteria:

* without previous orthodontic treatment, without systemic disesases and adenotonsillar hypertrophy.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children bewten 10-16 years old
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Impact of Twin Block and Motion Class II Appliances on Hyoid Bone Position - A Retrospective Clinical Study | 2023-2024
  See the impact of twin block and motion on the hyoid bone

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided